CLINICAL TRIAL: NCT01351623
Title: Phase II Study of Infusional Carfilzomib in Patients With Relapsed or Refractory Multiple Myeloma
Brief Title: Infusional Carfilzomib in Patients With Relapsed or Refractory Multiple Myeloma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10-228
Record Dates: First submitted 2011-05-09; First posted 2011-05-11 (Estimated); Results first posted 2017-03-13 (Actual); Last update posted 2017-04-13 (Actual); Status verified 2017-03

CONDITIONS: Multiple Myeloma
Keywords: PR-171 (CARFILZOMIB); Chemotherapy; 10-228
MeSH Terms: conditions — Multiple Myeloma | interventions — carfilzomib

ARMS (1):
- Carfilzomib (Experimental): A single arm, open-label, single institution phase 2 clinical trial is planned.
  Interventions: Drug: Carfilzomib

INTERVENTIONS:
Drug: Carfilzomib — Following enrollment patients will be treated with single agent infusional carfilzomib at 56mg/m2. Carfilzomib will be administered intravenously over 30 minutes on Days 1, 2, 8, 9, 15 and 16 of a 28-day cycle. Dexamethasone 8 mg PO/IV will be administered prior to all carfilzomib doses during the first cycle.

SUMMARY:
The purpose of this study is to test a new drug called carfilzomib. It is a type of drug called a proteasome inhibitor. Proteasome breaks down proteins that are no longer useful to the cell. When the proteasome is turned off by a drug (like carfilzomib), useless proteins cannot be broken down. Instead the proteins build up and cause the cell to die. Myeloma cells make a lot of protein and are especially in need of a functional proteasome to survive.

Carfilzomib is not approved for use by the Food and Drug Administration to treat myeloma. It is considered an experimental drug. Previous studies have shown that carfilzomib is safe to use. This study will look at what the effects, good and/or bad, carfilzomib has on myeloma.

ELIGIBILITY:
Inclusion Criteria:

* Participants must meet all of the following inclusion criteria to be eligible to enroll in this study.
* Patients meeting the criteria for symptomatic multiple myeloma that has relapsed or is refractory to at least 2 prior lines of therapy.
* Previous therapy with bortezomib.
* Previous therapy with thalidomide or lenalidomide.
* Patients must have measurable disease and therefore must have at least one of the following:

Serum M-protein ≥1 gm/dL (≥10 gm/L) Urine M-protein ≥200 mg/24 hr Serum FLC assay: involved FLC ≥10 mg/dL (≥100 mg/L) provided serum FLC ratio is abnormal.

* Age ≥ 18 years
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2 Adequate hepatic function, with serum ALT ≤ 3.5 times the upper limit of normal and serum direct bilirubin ≤ 2 mg/dL (34 µmol/L) within 14 days prior to enrollment
* Absolute neutrophil count (ANC) ≥ 1.0 × 109/L within 14 days prior to enrollment Hemoglobin ≥ 8 g/dL (80 g/L) within 14 days prior to enrollment (participants may be receiving red blood cell [RBC] transfusions in accordance with institutional guidelines)
* Platelet count ≥ 50 × 109/L (≥ 30 × 109/L if thought to be secondary to myeloma involvement of the bone marrow ) within 14 days prior to enrollment (platelet transfusions are allowed)
* Creatinine clearance (CrCl) ≥ 15 mL/minute within 14 days prior to enrollment, either estimated or calculated using a standard formula (eg, Cockcroft and Gault)
* Females of childbearing potential (FCBP) must agree to ongoing pregnancy testing and to practice contraception.
* Male participants must agree to practice contraception.

Exclusion Criteria:

* Prior treatment with carfilzomib.
* Known CNS involvement with myeloma
* Pregnant or lactating females
* Major surgery within 21 days prior to registration.
* Acute active infection requiring treatment (systemic antibiotics, antivirals, or antifungals) within 7 days prior to enrollment
* Known human immunodeficiency virus infection
* Active hepatitis B or C infection
* Unstable angina or myocardial infarction within 4 months prior to enrollment, NYHA Class III or IV heart failure, uncontrolled angina, severe uncontrolled ventricular arrhythmias, sick sinus syndrome, or electrocardiographic evidence of acute ischemia or Grade 3 conduction system abnormalities unless participant has a pacemaker
* Uncontrolled hypertension or uncontrolled diabetes within 14 days prior to enrollment.
* Concurrent malignancies, except for treated non-melanoma skin cancer and cervical carcinoma in situ.
* Significant neuropathy (Grades 3-4, ) within 14 days prior to enrollment
* Known history of allergy to Captisol® (a cyclodextrin derivative used to solubilize carfilzomib)
* Contraindication to any of the required concomitant drugs or supportive treatments, including options, antiviral drugs, or intolerance to hydration due to preexisting pulmonary or cardiac impairment
* Concurrent therapy with any other anticancer therapeutic with activity against multiple myeloma
* Concurrent therapy with investigative agents (e.g., antibiotics or antiemetics)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2011-05-09; Primary Completion 2016-01-26 (Actual); Study Completion 2016-01-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nikoletta Lendvai, MD,PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- [Derived] Lendvai N, Hilden P, Devlin S, Landau H, Hassoun H, Lesokhin AM, Tsakos I, Redling K, Koehne G, Chung DJ, Schaffer WL, Giralt SA. A phase 2 single-center study of carfilzomib 56 mg/m2 with or without low-dose dexamethasone in relapsed multiple myeloma. Blood. 2014 Aug 7;124(6):899-906. doi: 10.1182/blood-2014-02-556308. Epub 2014 Jun 24. PMID 24963043
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Carfilzomib
Started | 44
Completed | 35
Not Completed | 9
Not completed — Protocol Violation | 2
Not completed — Adverse Event | 4
Not completed — Withdrawal by Subject | 1
Not completed — Death | 2

BASELINE CHARACTERISTICS:
Arm/Group | Carfilzomib
Number analyzed (Participants) | 44
Age, Continuous [Median (Full Range); unit: years] | 63 [45 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25
  Male | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9
  Not Hispanic or Latino | 34
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 18
  White | 23
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 44

OUTCOME MEASURES:

1. Primary Outcome: To Evaluate the Best Overall Response Rate (ORR)
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI and/or CT: Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Stable Disease (SD), neither sufficient shrinkage to qualify for a Partial Response nor sufficient increase to qualify for Progression of Disease (POD); POD, 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions; Complete Response (CR), Disappearance of all target lesions
Time Frame: 2 years
Population: Participants who completed 4 cycles of treatment or whose disease progressed prior to completion of 4 cycles.
Measure: Count of Participants; unit: Participants
Arm/Group | Carfilzomib
Number analyzed (Participants) | 35
Participants
  Complete Response/CR | 1
  Very Good Partial Response/PR | 8
  Partial Response/PR | 9
  Minimal Response/MR | 3
  Stable Disease/SD | 2
  Progressin of Disease/POD | 12

ADVERSE EVENTS:
Arm/Group | Carfilzomib
Serious Adverse Events (participants affected / at risk) | 28/44
Other Adverse Events (participants affected / at risk) | 44/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Carfilzomib (N=44)
Abdominal Infection (Infections and infestations) | 1
Acute kidney injury (Renal and urinary disorders) | 4
Anemia (Blood and lymphatic system disorders) | 3
Appendicitis (Gastrointestinal disorders) | 1
Blood and lymphatic system disorders - Other, spec (Blood and lymphatic system disorders) | 2
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1
Chest pain - cardiac (Cardiac disorders) | 1
Confusion (Psychiatric disorders) | 1
Death NOS (Blood and lymphatic system disorders) | 4 — Participants expired due to progression of disease
Diarrhea (Gastrointestinal disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5
Febrile neutropenia (Blood and lymphatic system disorders) | 2
Heart failure (Cardiac disorders) | 3
Hypercalcemia (Blood and lymphatic system disorders) | 2
Hyperkalemia (Blood and lymphatic system disorders) | 2
Hypertension (Cardiac disorders) | 4
Hypotension (Cardiac disorders) | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2
Infections and infestations - Other (Infections and infestations) | 3
Intracranial hemorrhage (Blood and lymphatic system disorders) | 1
Lung infection (Respiratory, thoracic and mediastinal disorders) | 6
Myelodysplastic syndrome (Blood and lymphatic system disorders) | 1
Platelet count decreased (Blood and lymphatic system disorders) | 5
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 4
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3
Sepsis (Infections and infestations) | 2
Upper respiratory infection (Infections and infestations) | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Carfilzomib (N=44)
Diarrhea (Gastrointestinal disorders) | 29
Nausea (General disorders) | 26
Fatigue (General disorders) | 24
Headache (General disorders) | 23
Constipation (Gastrointestinal disorders) | 22
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 18
Peripheral edema (Cardiac disorders) | 17
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 16
Rash (Skin and subcutaneous tissue disorders) | 16
Arthralgia (General disorders) | 16
Hypertension (Cardiac disorders) | 12
Heart failure (Cardiac disorders) | 11
Lymphopenia (Blood and lymphatic system disorders) | 22
Leukopenia (Blood and lymphatic system disorders) | 19
Thrombocytopenia (Blood and lymphatic system disorders) | 17
Anemia (Blood and lymphatic system disorders) | 16
Neutropenia (Blood and lymphatic system disorders) | 10
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 8
Hypophosphatemia (Blood and lymphatic system disorders) | 7
Hyponatremia (Blood and lymphatic system disorders) | 5
Hypocalcemia (Blood and lymphatic system disorders) | 5
ALT increased (Hepatobiliary disorders) | 3
AST increased (Hepatobiliary disorders) | 3
Hyperglycemia (Metabolism and nutrition disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes